CLINICAL TRIAL: NCT00477542
Title: A Phase I Trial of Myeloablative Conditioning Using Clofarabine and High-Dose Busulfan for Patients With Refractory Hematological Malignancies Undergoing Allogeneic HSCT
Brief Title: A Phase I Trial of Myeloablative Conditioning w/ Clofarabine and HD Busulfan for Pts w/ Refractory Heme Malignancies Undergoing Allo PBSCT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0704-30 IUCRO-0186
Record Dates: First submitted 2007-05-21; First posted 2007-05-23 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Hematologic Malignancies
Keywords: Clofarabine; allogeneic HSCT; refractory malignancies
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: clofarabine — Cohort- n- Clofarabine (mg/m2/day)
  -1 3-10 20
  1. 3-6 30
  2. 3-6 40
  3. 3-6 50
  4. 3-6 60
  5. 6-10 70

SUMMARY:
This is a phase trial to determine the maximum tolerated dose (MTD) of clofarabine in a combination with a myeloablative dose of busulfan. This is an initial step in developing a novel myeloablative preparative regimen for allogeneic hematopoietic stem cell transplantation (HSCT). While this phase I trial will initially develop the regimen in patients with refractory disease, it is expected that it will find its best application in patients with less advanced disease

DETAILED DESCRIPTION:
All patients will receive the same dose of busulfan. The dose of clofarabine will be escalated in successive cohorts of patients. Using a standard dose escalation design, successive cohorts of 3 patients will be treated with escalating doses of clofarabine. At the MTD (or highest dose-level if the MTD is not reached), the cohort will be expanded to 10 patients to better investigate correlative studies and give some preliminary idea of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of disease. Patients must have one of the following disease types:

  * Acute myeloid leukemia (AML) with either:

    * Primary refractory to induction chemotherapy
    * Relapsed and refractory AML with >5% blasts in bone marrow or extramedullary disease (excluding active disease of the central nervous system).
    * Patients in second or subsequent complete remission (CR2, CR3, etc.).
  * Acute lymphoblastic leukemia (ALL) with one of the following criteria:

    * Primary refractory to induction chemotherapy.
    * Relapsed and refractory ALL with >5% blasts in bone marrow or extramedullary disease (excluding active disease of the central nervous system).
    * Patients in second or subsequent complete remission (CR2, CR3, etc.).
  * Myelodysplasia, refractory anemia with excess blasts with 11-20% blasts in the bone marrow (RAEB II).
  * Chronic myelogenous leukemia (CML) with one of the following criteria:

    * Accelerated phase.
    * Patients in blast crisis.
  * Patients with aggressive non-Hodgkin's lymphoma (NHL), including diffuse large cell lymphoma, mediastinal B-cell lymphoma, transformed lymphoma, mantle cell lymphoma, and peripheral T cell lymphoma, who also have one of the following criteria:

    * Failure to achieve complete remission to primary induction therapy
    * Relapsed NHL, refractory to at least one line of salvage systemic therapy
* Patients who relapse < 6 months following autologous stem cell transplantation are not eligible.
* Patient age 18-60 years
* Availability of a consenting HLA-matched donor
* Performance status ECOG 0-1
* No active infection. Patients with active infections requiring oral or intravenous antibiotics are not eligible for enrollment until resolution of infection.
* No HIV disease. Patients with immune dysfunction are at a significantly higher risk of infection from intensive immunosuppressive therapies.
* Non-pregnant and non-nursing. Treatment under this protocol would expose a fetus to significant risks. Women of childbearing potential should have a negative pregnancy test prior to study entry. Women and men of reproductive potential should agree to use an appropriate method of birth control throughout their participation in this study due to the teratogenic potential of the therapy utilized in this trial. Appropriate methods of birth control include oral contraceptives, implantable hormonal contraceptives (Norplant®), or double barrier method (diaphragm plus condom).
* Required baseline laboratory values:

  * LVEF > 45% corrected
  * DLCO > 50% of predicted value (corrected for hemoglobin)
  * Serum creatinine ≤ 2.0 mg/dl or estimated creatinine clearance of ≥60 ml/min
  * Bilirubin < 1 x upper limit of normal value
  * AST and ALT < 1 x upper limit of normal value
* Signed written informed consent. Patient must be capable of understanding the investigational nature of the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent.

Exclusion Criteria:

* Patients who relapse < 6 months following autologous stem cell transplantation are not eligible

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Determine the MTD of clofarabine in association with a myeloablative dose of busulfan as a preparative regimen in patients with refractory hematological malignancies undergoing allogeneic HSCT. | 1 year

SECONDARY OUTCOMES:
• Assessment of the toxicity of the combination of clofarabine and busulfan • Assess clofarabine and busulfan pharmacokinetics with combination therapy • Describe the response rate • Describe relapse rate and event-free survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Farag, MD, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States